CLINICAL TRIAL: NCT03046927
Title: Vitamin D and Residual Beta-Cell Function in Type 1 Diabetes
Acronym: PCR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benjamin U. Nwosu, MD (Other)
Collaborators: University of Massachusetts, Worcester (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Benjamin U. Nwosu, MD, Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H00010550; 1R21DK113353 (NIH)
Record Dates: First submitted 2017-02-01; First posted 2017-02-08 (Estimated); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; vitamin D; honeymoon phase
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Ergocalciferols; Vitamin D

STUDY DESIGN:
Intervention Model Description: 12-month randomized, double-blind, placebo-controlled, parallel design trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Ergocalciferol and placebo will be prepared as identical capsules by Boulevard Pharmaceutical Compounding Center. Randomization will be conducted by the Investigational Drug Services (IDS), UMMS, using a randomization scheme generated by Dr. Barton. Randomization will be 1:1 (ergocalciferol: placebo) and will use a permuted block design with blocking for every 2 or 4 subjects (at random). IDS will maintain blinding information and PI will contact IDS for emergency unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ergocalciferol (Experimental): Oral administration of 50,000 IU of ergocalciferol one capsule per week for 2 months; and then once every 2 weeks for 10 months in 20 subjects of 10-21yr with newly diagnosed T1D
  Interventions: Drug: Ergocalciferol
- Placebo (Placebo Comparator): Oral administration of placebo one capsule per week for 2 months; and then once every 2 weeks for 10 months in 20 subjects of 10-21yr with newly diagnosed T1D
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ergocalciferol — Each subject on the experimental arm will receive one capsule of ergocalciferol per week for 2 months; and then once every 2 weeks for 10 months
  Other Names: Vitamin D
  Arms: Ergocalciferol
Other: Placebo — Each subject on the placebo arm will receive one capsule of placebo per week for 2 months; and then once every 2 weeks for 10 months
  Arms: Placebo

SUMMARY:
This project is designed to study the role of vitamin D supplementation on the honeymoon phase of type 1 diabetes in children who are on standardized insulin treatment. The results could lead to significant changes in the approach to the early phase of type 1 diabetes with a strong emphasis on prolonging the honeymoon phase by using vitamin D and maintaining these patients on a standardized insulin regimen. The overall goal is to reduce the long-term complications of type 1 diabetes.

DETAILED DESCRIPTION:
Prolonging the duration of the partial clinical remission (PCR), or 'honeymoon' phase, of type 1 diabetes (T1D) improves glycemic control and reduces long-term complications. Recent studies suggest the exciting possibility that vitamin D supplementation, a safe and easy-to-implement therapy in children, may lengthen PCR and increase residual beta cell function (RBCF).

However, existing studies employed a suboptimal vitamin D dose or lacked a standardized insulin treatment protocol, precluding solid conclusions and preventing the field from moving forward with translation to clinical practice. This trial's rationale is to securely establish the effect of an adequate dose of vitamin D on PCR and RBCF.

We hypothesize that vitamin D will increase RBCF and prolong PCR. The primary aim is to determine the effect of adjunctive vitamin D on RBCF and PCR in youth with T1D maintained on a standardized insulin protocol. We propose a 12-month randomized, double-blind, placebo-controlled, parallel design trial of ergocalciferol vs. placebo in 40 subjects of 10-21 years with newly-diagnosed T1D. The primary outcome is the change over time in stimulated C-peptide (a measure of RBCF). Secondary outcomes include change over time in insulin-dose-adjusted-hemoglobin-A1c (HbA1c) (IDAA1C; a measure of PCR), HbA1c, and total daily dose of insulin. Mechanistic studies will explore whether beneficial effects of vitamin D are associated with increased GLP-1 levels or decreased inflammatory markers, and whether response to vitamin D is impacted by T1D-risk polymorphisms. If our hypotheses are true, these findings may completely alter the approach to the early management of T1D, with strong emphasis on prolonging the honeymoon phase using a readily available and easily affordable vitamin D while maintaining these patients on a standardized insulin treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 10-21 years.
2. Sex: male and female subjects will be enrolled.
3. Tanner stage: I-V.
4. T1D duration of <3 months (i.e., from first insulin injection) to ensure the inclusion of patients in PCR.
5. Presence of at least one diabetes-associated autoantibody.
6. Normal-weight, overweight-, and obese subjects with T1D
7. Fasting serum C-peptide level of >0.1 nmol/L (0.3 ng/mL)1; or 2-hour post-meal stimulated C-peptide level of 0.2 nmol/L (≥0.6 ng/mL).

Exclusion Criteria:

1. Subjects on weight altering medications, such as orlistat.
2. Subjects with eating disorders
3. Subjects on medications other than insulin that can affect blood glucose level.
4. Subjects with 25-hydroxyvitamin D [25(OH)D] levels of >70 ng/mL, as this may lead to vitamin D toxicity in the study subjects.
5. Subjects with systemic diseases other than T1D.
6. Subjects with recurrent diabetic ketoacidosis (>2 episodes since the diagnosis of T1D or in the preceding 3 months); or >2 episodes of severe hypoglycemia in the preceding 3 mo.
7. Pregnant or breast-feeding female subjects.
8. The receipt of any investigational drug within 6 months prior to this trial.
9. Active malignant neoplasm.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin U Nwosu, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 48 enrolled participants, 36 met the inclusion criteria and were randomized to the treatment.
Period: Overall Study
Arm/Group | Ergocalciferol | Placebo
Started | 18 | 18
Completed | 13 | 16
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ergocalciferol | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.25 (2.76) | 14.28 (2.86) | 13.77 (2.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 10 | 14 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
HbA1C [Mean (Standard Deviation); unit: Percentage of HbA1C] | 7.62 (1.35) | 7.47 (1.69) | 7.54 (1.52)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 22.03 (5.41) | 22.01 (4.15) | 22.02 (4.73)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dl] | 125.83 (25) | 111.13 (35.78) | 118.91 (30.97)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 76.16 (14.83) | 76.22 (11.56) | 76.19 (13.14)
Height [Mean (Standard Deviation); unit: cm] | 156.12 (12.77) | 158.65 (11.30) | 157.38 (11.96)
Height Z-score [Mean (Standard Deviation); unit: Z-score] — A z-score is the same as standard deviation score; A height z-score of 0 represents the population mean; A z-score above the mean is considered better than a z-score below the mean; A height z-score of >2 indicates tall stature, while a height z-score <2 indicates short stature
  Z-score | 0.50 (0.73) | 0.48 (1.18) | 0.49 (0.96)
weight [Mean (Standard Deviation); unit: kg] | 53.33 (15.19) | 56.16 (14.66) | 54.78 (14.77)
Weight z-score [Mean (Standard Deviation); unit: Z-score] — A z-score is the same as standard deviation score; A weight z-score of 0 represents the population mean; A weight z-score below the mean is considered better than a z-score above the mean; A weight z-score of >2 indicates overweight/obesity, while a weight z-score <2 indicates underweight
  Z-score | 0.86 (0.81) | 0.67 (0.68) | 0.76 (0.74)
Body mass index z-score [Mean (Standard Deviation); unit: Z-score] — A z-score is the same as standard deviation score; A BMI z-score of 0 represents the population mean; A BMI z-score below the mean is considered better than a BMI z-score above the mean; A BMI z-score of >2 indicates overweight/obesity, while a weight z-score <2 indicates underweight
  Z-score | 0.89 (0.94) | 0.74 (0.68) | 0.82 (0.81)
systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 104.94 (9.06) | 106.44 (10.60) | 105.69 (9.74)
diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 64.72 (9.14) | 64.67 (6.80) | 64.69 (7.94)
Total Daily Dose (TDD) Insulin [Mean (Standard Deviation); unit: units/d] | 37 (29.61) | 27.17 (14.41) | 31.94 (23.27)
Total Daily Dose Insulin [Mean (Standard Deviation); unit: units/kg/d] | 0.51 (0.23) | 0.48 (0.23) | 0.50 (0.23)
Total Daily Dose Long-acting insulin only [Mean (Standard Deviation); unit: units] | 18.50 (14.81) | 14.14 (7.30) | 16.26 (11.60)
puberty stage, tanner II-V [Count of Participants; unit: Participants] | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Residual Beta-cell Function (RBCF)
Description: Investigation of the effect of vitamin D on residual beta cell function (RBCF) in the first 12 months after the diagnosis of T1D by using stimulated C-peptide levels to quantify RBCF.
Time Frame: Baseline to 12 months at 3 months interval
Population: individuals aged 10-21 years with newly diagnosed T1D in a 12-month RCT of ergocalciferol vs placebo to determine the effect of vitamin D on RBCF and PR in youth with newly diagnosed T1D.
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Ergocalciferol | Placebo
Number analyzed (Participants) | 18 | 18
ng/ml
  Baseline | 1.78 (0.28) | 2.27 (0.31)
  Mo 3 | 1.56 (0.25) | 1.76 (0.21)
  Mo 6 | 1.40 (0.26) | 1.53 (0.25)
  Mo 9 | 1.25 (0.24) | 1.36 (0.31)
  Mo 12 | 1.05 (0.22) | 1.15 (0.29)
Statistical Analysis 1: Comparison: Ergocalciferol vs Placebo; Test type: Equivalence — p values were obtained using generalized linear model with GEE for repeated measures; p < 0.001, generalized linear model with dependent; Mean Difference (Net) = 0.08 — Trend analysis was performed using generalized linear model with GEE for repeated measures

2. Secondary Outcome: Change in Percent of HbA1c From Baseline Over Time During Partial Clinical Remission (PCR)
Description: Effect of vitamin D supplementation on glycemic control during the partial clinical remission phase as shown by the change in percent HbA1c from baseline across longitudinal measurements at 0, 3, 6, 9, and 12 months.
Time Frame: Baseline to 12 months
Measure: Least Squares Mean (Standard Error); unit: percent of HbA1C
Arm/Group | Ergocalciferol | Placebo
Number analyzed (Participants) | 18 | 18
percent of HbA1C
  Baseline | 7.62 (0.32) | 7.47 (0.39)
  Mo 3 | 7.25 (0.37) | 6.67 (0.28)
  Mo 6 | 7.28 (0.27) | 7.15 (0.34)
  Mo 9 | 7.48 (0.35) | 7.61 (0.32)
  Mo 12 | 7.65 (0.57) | 8.03 (0.41)
Statistical Analysis 1: Comparison: Ergocalciferol vs Placebo; Test type: Other; p < 0.01, generalized linear model — The threshold for statistical significance was p=0.05; p values were obtained using generalized linear model with GEE for repeated measures; trend analysis = 0.04 — Trend analysis was performed using generalized linear model with GEE for repeated measures

3. Secondary Outcome: Glucagon-like Peptide-1 (GLP-1)
Description: Investigation of the effect of vitamin D supplementation on GLP-1 during PCR.
Time Frame: Baseline to 12 months at 3 months interval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Ergocalciferol | Placebo
Number analyzed (Participants) | 18 | 18
ng/ml
  Baseline | 10.26 (7.54) | 5.81 (3.38)
  Mo 3 | 8.58 (5.02) | 8.4 (5.48)
  Mo 6 | 10.24 (5.69) | 6.86 (3.01)
  Mo 9 | 10.26 (5.57) | 8.89 (5.69)
  Mo 12 | 9.11 (4.44) | 9.63 (5.92)
Statistical Analysis 1: Comparison: Ergocalciferol vs Placebo; Test type: Other — p values were derived from trend analysis using generalized linear models; p = 0.0241, General linear models — The p-value was derived from a statistical model adjusted for age, sex, and BMI; Mean Difference (Net) = 0.507, 95% CI 2-sided [0.066 to 0.947]

4. Secondary Outcome: Vitamin D Binding Protein (VDBP)
Description: Investigation of the effect of vitamin D supplementation on VDBP during PCR.
Time Frame: Baseline to 12 months at 3 months interval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Ergocalciferol | Placebo
Number analyzed (Participants) | 18 | 18
ng/ml
  Baseline | 134.32 (22.82) | 111.56 (28.82)
  Mo 3 | 118.11 (27.93) | 118.79 (22.96)
  Mo 6 | 135.32 (27.51) | 138.18 (33.15)
  Mo 9 | 135.79 (38.47) | 131.51 (38.86)
  Mo 12 | 141.34 (32.8) | 152.42 (31.19)
Statistical Analysis 1: Comparison: Ergocalciferol vs Placebo; Test type: Other — p values were obtained from a generalized linear model with repeated measures; p = 0.23, Regression, Linear — The p-value was derived from a statistical model adjusted for age, sex, and BMI; Mean Difference (Net) = 10.37, 95% CI 2-sided [-6.40 to 27.13]

5. Secondary Outcome: Effect of Vitamin D Supplementation on the Duration of Partial Clinical Remission (PCR) of Type 1 Diabetes
Description: Insulin dose-adjusted hemoglobin A1c (HbA1c) (IDAA1C)
Time Frame: Baseline to12 months 3 monthly
Population: individuals aged 10 to 21 years with newly diagnosed T1D in a 12-month RCT of ergocalciferol vs placebo to determine the effect of vitamin D on RBCF and PR in youth with newly diagnosed T1D.
Measure: Least Squares Mean (Standard Error); unit: % of IDAA1c
Arm/Group | Ergocalciferol | Placebo
Number analyzed (Participants) | 18 | 18
% of IDAA1c
  Baseline | 9.9 (0.4) | 9.4 (0.6)
  Mo 3 | 9.7 (0.6) | 8.4 (0.4)
  Mo 6 | 10.0 (0.5) | 9 (0.5)
  Mo 9 | 10.4 (0.5) | 10.1 (0.5)
  Mo 12 | 10.6 (0.6) | 10.7 (0.6)
Statistical Analysis 1: Comparison: Ergocalciferol vs Placebo; Test type: Other; p < 0.001, generalized linear model; p values were obtained using generalized linear model with GEE for repeated measures; trend analysis = .02; Trend analysis was obtained using generalized linear model GEE

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Ergocalciferol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 7/18 | 3/18
Other Adverse Events (participants affected / at risk) | 1/18 | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ergocalciferol (N=18) | Placebo (N=18)
Diabetic ketoacidosis (Endocrine disorders) | 0 | 1
Hyperglycemia (Endocrine disorders) | 3 | 1
mild hypoglycemia (Endocrine disorders) | 3 | 1
moderate hypoglycemia (Endocrine disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ergocalciferol (N=18) | Placebo (N=18)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 5
mild hair loss (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT03046927/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT03046927/SAP_001.pdf